CLINICAL TRIAL: NCT02651350
Title: A Randomized Controlled Clinical Trial on the Efficacy and Safety of Glucocorticosteroid in the Patients With Chronic Recurrent Drug-induced Liver Injury
Brief Title: Efficacy and Safety of Glucocorticosteroid Treatment in the Patients With Chronic Recurrent DILI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJ302-FGRXGB-001
Record Dates: First submitted 2015-12-25; First posted 2016-01-11 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2019-07

CONDITIONS: Drug-induced Liver Injury,Chronic
Keywords: Drug-induced Liver Injury; Recurrence; Methylprednisolone
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury, Chronic; Chemical and Drug Induced Liver Injury; Recurrence | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone (Experimental): Participants will receive methylprednisolone from week 0 through week 48 study visit in combination with standard treatment including reduced glutathione, glycyrrhizin, ademetionine, alprostadil,or ursodeoxycholic acid (UDCA) in the first 12 weeks. Participants will then be followed until week 72 study visit.
  Interventions: Drug: Methylprednisolone; Drug: Standard Treatment
- Standard Treatment (Active Comparator): Participants will only receive standard treatment (namely,routine liver protection drugs) including reduced glutathione, glycyrrhizin, ademetionine, alprostadil,or ursodeoxycholic acid (UDCA) from week 0 through week 12 study visit. Participants will then be followed until week 72 study visit.
  Interventions: Drug: Standard Treatment

INTERVENTIONS:
Drug: Methylprednisolone — Participants will receive methylprednisolone,48mg/d for the 1st week,32mg/d for the 2nd week,24mg/d for the next two weeks, followed by 16mg/d for 32 weeks and reduction in doses of methylprednisolone by 4 mg per 4 weeks until drug withdrawal.Participants will also receive standard treatment including reduced glutathione, glycyrrhizin, ademetionine, alprostadil, or ursodeoxycholic acid (UDCA) in the first 12 weeks.The total treatment duration will be 48 weeks. Follow-up duration is 24 weeks.
  Other Names: MEDROL,NDC0009-0056-02
  Arms: Methylprednisolone
Drug: Standard Treatment — Participants will only receive standard treatment,namely,routine liver protection drugs including reduced glutathione, glycyrrhizin, ademetionine, alprostadil,or ursodeoxycholic acid (UDCA) from week 0 through week 12 study visit. Participants will then be followed until week 72.
  Other Names: Routine liver protection drugs

SUMMARY:
This study is to observe the efficacy and safety of glucocorticosteroid treatment in the patients with chronic recurrent drug-induced liver injury (DILI).

DETAILED DESCRIPTION:
Drug-induced liver injury (DILI) refers to liver diseases caused by drugs and toxic substances. DILI is a clinical event that can be associated with severe outcomes such as acute liver failure. Up to now, approximately 1000 drugs, herbal products, vitamins and illicit compounds are associated with liver injury. Recently, the incidence of DILI is rising. In our hospital, hospitalized patients with DILI was increased from 1.39% in 2002 to 2.31% in 2006, and further up to 3.17% in 2011, which indicated 2.3-folds increase over last ten years.15% to 20% patients with acute DILI are prone to chronic liver disease. For patients with chronic recurrent DILI, routine liver protective treatment was difficult to rescue abnormal liver functions. Moreover, increasing health care costs seriously affect the patient's quality of life. Glucocorticosteroids can inhibit the non-specific inflammation and permeability of the capillary bile duct, limit the activation of T lymphocytes, and selectively inhibit B lymphocytes to produce antibodies, thus preventing or delaying the immune-induced liver injury. Glucocorticoid treatment of severe DILI has accepted some recognition, but the effect of repeated episodes of chronic DILI, due to a lack of randomized controlled studies, is still unclear. Therefore, we shall design two groups on the basis of the ratio of 1:1, namely, glucocorticoid treatment group and standard treatment alone group. Participants in glucocorticoid treatment group will receive methylprednisolone,48mg/d for the 1st week, 32mg/d for the 2nd week, 24mg/d for the next two weeks, followed by 16mg/d for 32 weeks and reduction in doses of methylprednisolone by 4 mg per 4 weeks until drug withdrawal. Participants in glucocorticoid treatment group also receive standard treatment including reduced glutathione, glycyrrhizin, ademetionine, alprostadil,or ursodeoxycholic acid (UDCA) in the first 12 weeks. Participants in standard treatment group will only receive treatment by routine liver protection drugs including reduced glutathione, glycyrrhizin, ademetionine, alprostadil, or ursodeoxycholic acid (UDCA) in the first 12 weeks.The efficacy and safety of glucocorticoid treatment in the patients with chronic recurrent DILI will be observed during the treatment and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Meet with ACG clinic guidelines for diagnostic criteria of chronic DILI;
2. Meet any of the following conditions:

   * serum AST or ALT ≥ 10 fold ULN;
   * serum AST or ALT ≥ 5 fold ULN and TBIL ≥ 2 fold ULN;
   * liver histology indicates bridging necrosis or multiacinar necrosis or moderate or more inflammation or inflammation G3 or more;
3. Women of childbearing age had a negative urine pregnancy test, and the subjects are willing to have no family planning during the study and to take effective measures;
4. Voluntary participation, understanding and signing of informed consent, comply with the requirements of the research;

Exclusion Criteria:

1. Patients with serious pre-existent comorbid conditions (vertebral compression fractures,psychosis,active peptic ulcer, brittle diabetes,uncontrolled hypertension;
2. Patients with intolerances to prednisone;
3. Patients with severe infection receiving antibiotics, anti-fungal,anti-viral therapy;
4. Viral hepatitis,alcoholic or non-alcoholic liver disease,Wilson's disease or other inherited metabolic liver diseases.
5. Pregnancy or desire of pregnancy;
6. Breast-feeding;
7. Liver cancer or other malignant tumor;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-12; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
The relapse or recurrent rate of illness, namely, appearance of obviously abnormal liver function again during treatment and follow-up period | At week 24
  The biochemical relapse rate was analyzed by either intention to treat (ITT) or per protocol set (PPS). Biochemical relapse was characterized either by the serum alanine transaminase (ALT) or aspartate aminotransferase (AST) ≥ 3 × upper limits of normal (ULN) or alkaline phosphatase (ALP) ≥ 2 × ULN, or by at least 2 folds increase in serum ALT or AST or ALP from the abnormal index lately.
The relapse or recurrent rate of illness, namely, appearance of obviously abnormal liver function again during treatment and follow-up period | At week 72
  The biochemical relapse rate was analyzed by either intention to treat (ITT) or per protocol set (PPS). Biochemical relapse was characterized either by the serum alanine transaminase (ALT) or aspartate aminotransferase (AST) ≥ 3 × upper limits of normal (ULN) or alkaline phosphatase (ALP) ≥ 2 × ULN, or by at least 2 folds increase in serum ALT or AST or ALP from the abnormal index lately.

SECONDARY OUTCOMES:
Days of normalization of liver functions including serum levels of ALT, AST, TBIL,GGT and ALP. | From week 1 to week 12
  The normalization time(days) of biochemistry was defined as the days of normalization of each biochemical parameter (ALT, AST, TBil, ALP and gamma-glutamyl transpeptidase), respectively.
The liver histological changes between two liver biopsies | At week 0 and at week 48 week
  Histological improvement was defined as at least two points reduce in the activity score, or at least one point decrease in the fibrosis score in accordance to Ishak scoring system.
The number of participants with methylprednisolone treatment-related adverse events, such as severe osteopenia, uncontrolled hypertension | At week 24 and at week 72
  The adverse effects in each group were evaluated according to the Common Terminology Criteria for Adverse Events (version 5.0). The types of steroid-related adverse effects referred to the EASL/AASLD autoimmune hepatitis Guidelines. Adverse effects occurred in both the treatment period and the follow-up period were combined to evaluate.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengsheng Zou, Dr., Principal Investigator — Beijing 302 Hospital,China.
Locations (1):
- Beijing 302 hospital,China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chalasani NP, Hayashi PH, Bonkovsky HL, Navarro VJ, Lee WM, Fontana RJ; Practice Parameters Committee of the American College of Gastroenterology. ACG Clinical Guideline: the diagnosis and management of idiosyncratic drug-induced liver injury. Am J Gastroenterol. 2014 Jul;109(7):950-66; quiz 967. doi: 10.1038/ajg.2014.131. Epub 2014 Jun 17. PMID 24935270
- [Background] Moreno L, Sanchez-Delgado J, Vergara M, Casas M, Miquel M, Dalmau B. Recurrent drug-induced liver injury (DILI) with ciprofloxacin and amoxicillin/clavulanic. Rev Esp Enferm Dig. 2015 Dec;107(12):767-8. doi: 10.17235/reed.2015.3810/2015. PMID 26671593
- [Background] Tencate V, Komorowski R, Cronin D, Hong J, Gawrieh S. A case study: refractory recurrent autoimmune hepatitis following liver transplantation in two male patients. Transplant Proc. 2014 Jan-Feb;46(1):298-300. doi: 10.1016/j.transproceed.2013.09.028. PMID 24507072
- [Background] Lucena MI, Kaplowitz N, Hallal H, Castiella A, Garcia-Bengoechea M, Otazua P, Berenguer M, Fernandez MC, Planas R, Andrade RJ. Recurrent drug-induced liver injury (DILI) with different drugs in the Spanish Registry: the dilemma of the relationship to autoimmune hepatitis. J Hepatol. 2011 Oct;55(4):820-7. doi: 10.1016/j.jhep.2010.12.041. Epub 2011 Feb 19. PMID 21338638
- [Background] Suzuki A, Brunt EM, Kleiner DE, Miquel R, Smyrk TC, Andrade RJ, Lucena MI, Castiella A, Lindor K, Bjornsson E. The use of liver biopsy evaluation in discrimination of idiopathic autoimmune hepatitis versus drug-induced liver injury. Hepatology. 2011 Sep 2;54(3):931-9. doi: 10.1002/hep.24481. Epub 2011 Aug 8. PMID 21674554
- [Background] Weiler-Normann C, Schramm C. Drug induced liver injury and its relationship to autoimmune hepatitis. J Hepatol. 2011 Oct;55(4):747-9. doi: 10.1016/j.jhep.2011.02.024. Epub 2011 Mar 9. No abstract available. PMID 21396413
- [Background] Bessone F, Lucena MI, Roma MG, Stephens C, Medina-Caliz I, Frider B, Tsariktsian G, Hernandez N, Bruguera M, Gualano G, Fassio E, Montero J, Reggiardo MV, Ferretti S, Colombato L, Tanno F, Ferrer J, Zeno L, Tanno H, Andrade RJ. Cyproterone acetate induces a wide spectrum of acute liver damage including corticosteroid-responsive hepatitis: report of 22 cases. Liver Int. 2016 Feb;36(2):302-10. doi: 10.1111/liv.12899. Epub 2015 Jul 16. PMID 26104271
- [Background] Sugimoto K, Ito T, Yamamoto N, Shiraki K. Seven cases of autoimmune hepatitis that developed after drug-induced liver injury. Hepatology. 2011 Nov;54(5):1892-3. doi: 10.1002/hep.24513. Epub 2011 Aug 9. No abstract available. PMID 21725992
- [Background] Fujiwara K, Yokosuka O. Histological discrimination between autoimmune hepatitis and drug-induced liver injury. Hepatology. 2012 Feb;55(2):657. doi: 10.1002/hep.24768. No abstract available. PMID 22038865
- [Background] Manns MP, Czaja AJ, Gorham JD, Krawitt EL, Mieli-Vergani G, Vergani D, Vierling JM; American Association for the Study of Liver Diseases. Diagnosis and management of autoimmune hepatitis. Hepatology. 2010 Jun;51(6):2193-213. doi: 10.1002/hep.23584. No abstract available. PMID 20513004
- [Background] Fontana RJ, Hayashi PH, Gu J, Reddy KR, Barnhart H, Watkins PB, Serrano J, Lee WM, Chalasani N, Stolz A, Davern T, Talwakar JA; DILIN Network. Idiosyncratic drug-induced liver injury is associated with substantial morbidity and mortality within 6 months from onset. Gastroenterology. 2014 Jul;147(1):96-108.e4. doi: 10.1053/j.gastro.2014.03.045. Epub 2014 Mar 27. PMID 24681128
- [Derived] Wang JB, Huang A, Wang Y, Ji D, Liang QS, Zhao J, Zhou G, Liu S, Niu M, Sun Y, Tian H, Teng GJ, Chang BX, Bi JF, Peng XX, Xin S, Xie H, Ma X, Mao YM, Liangpunsakul S, Saxena R, Aithal GP, Xiao XH, Zhao J, Zou Z. Corticosteroid plus glycyrrhizin therapy for chronic drug- or herb-induced liver injury achieves biochemical and histological improvements: a randomised open-label trial. Aliment Pharmacol Ther. 2022 May;55(10):1297-1310. doi: 10.1111/apt.16902. Epub 2022 Mar 31. PMID 35362188